CLINICAL TRIAL: NCT02054702
Title: Protocol 331-13-008: An Exploratory, Multicenter, Open-label, Flexible-dose Brexpiprazole (OPC-34712) Trial in Adults With Acute Schizophrenia
Brief Title: Brexpiprazole (OPC-34712) Trial in the Treatment of Adults With Acute Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 331-13-008
Record Dates: First submitted 2014-02-02; First posted 2014-02-04 (Estimated); Results first posted 2015-12-01 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mental Disorders; Psychotic Disorders; Antipsychotic; Cognitive testing
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders | interventions — brexpiprazole; Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brexpiprazole (Experimental): Treatment (6 weeks) Up to 4 mg/day, once daily dose, tablets, orally
  Interventions: Drug: Brexpiprazole
- Aripiprazole (Experimental): Aripiprazole - Up to 20 mg/day, once daily dose, tablets, orally
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Treatment (6 weeks) Up to 4 mg/day, once daily dose, tablets, orally
  Arms: Brexpiprazole
Drug: Aripiprazole — Up to 20 mg/day, once daily dose, tablets, orally
  Arms: Aripiprazole

SUMMARY:
The purpose of this study is to explore changes in efficacy, cognitive functioning, and safety of flexibly-dosed Brexpiprazole monotherapy in subjects with acute schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age, inclusive, at the time of informed consent with a diagnosis of schizophrenia as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I) for Schizophrenia and Psychotic Disorders Studies
* Would benefit from hospitalization or continued hospitalization for treatment of a current acute relapse of schizophrenia at trial entry
* Are experiencing an acute exacerbation of psychotic symptoms and marked deterioration of usual function as demonstrated by all of the following:
* Positive and Negative Syndrome Scale (PANSS) Total Score of ≥ 80
* Score of ≥ 4 on two or more of the following PANSS items at screening: hallucinatory behavior, unusual thought content, conceptual disorganization, or suspiciousness
* Clinical Global Impression - Severity of Illness Scale (CGI-S) score ≥ 4 (moderately ill)

Exclusion Criteria:

* Are presenting with a first episode of schizophrenia based on the clinical judgment of the investigator
* Have been hospitalized > 21 days for the current acute episode at the time of the baseline visit
* Have a current DSM-IV-TR Axis I diagnosis other than schizophrenia, including, but not limited to, schizoaffective disorder, major depressive disorder (MDD), bipolar disorder, post-traumatic stress disorder, anxiety disorders, delirium, dementia, amnestic, or other cognitive disorders; also borderline, paranoid, histrionic, schizotypal, schizoid, antisocial personality disorders or mental retardation.
* Improvement of ≥ 20% in total PANSS score between the screening and baseline assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd Japan (OPCJ)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 97 participants at 19 trial sites in United States.
Pre-assignment Details: The trial consisted of a 2- to 14-day screening phase, a 6-week treatment phase, and a 30-day follow-up phase.
Groups:
- Brexpiprazole: Participants were administered brexpiprazole tablets orally, once daily (QD) starting dose at 1 milligram per day (mg/day) for 4 days followed by 2 mg/day for 3 days and 3 mg/day at the week 1 visit and 1, 2, 3, or 4 mg/day from week 2 to week 6.
- Aripiprazole: Participants were administered aripiprazole tablets orally QD, starting dose at 10 mg/day for 1 week, followed by 15 mg/day at the Week 1 visit and 10, 15, or 20 mg/day from week 2 to week 6.
Period: Overall Study
Arm/Group | Brexpiprazole | Aripiprazole
Started | 64 | 33
Completed | 40 | 21
Not Completed | 24 | 12
Not completed — Lost to Follow-up | 3 | 5
Not completed — Adverse Event | 3 | 1
Not completed — Met Withdrawal Criteria | 4 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 14 | 4

BASELINE CHARACTERISTICS:
Groups:
- Brexpiprazole: Participants were administered brexpiprazole tablets orally QD, starting dose at 1 mg/day for 4 days followed by 2 mg/day for 3 days and 3 mg/day at the week 1 visit and 1, 2, 3, or 4 mg/day from week 2 to week 6.
- Arpiprazole: Participants were administered aripiprazole tablets orally QD, starting dose at 10 mg/day for 1 week, followed by 15 mg/day at the Week 1 visit and 10, 15, or 20 mg/day from week 2 to week 6.
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole | Arpiprazole | Total
Number analyzed (Participants) | 64 | 33 | 97
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.2 (10.1) | 42.1 (10.4) | 42.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 46 | 23 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome).
Time Frame: Baseline to Week 6
Population: All randomized participants who took at least one dose of study medication and who had a valid Baseline assessment and at least 1 valid Post-Baseline efficacy assessment. The efficacy analyses were performed by fitting a mixed model repeated measures (MMRM) analysis with an unstructured variance covariance structure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
Units on a scale | -22.9 (1.7) | -19.4 (2.4)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in PANSS total score from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in PANSS total score from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

2. Secondary Outcome: Change From Baseline in Cognitive Test Battery Composite Score
Description: The cognitive test battery contains 8-tasks, including the Detection Task (DET, speed of processing), Identification Task (IDN, attention/vigilance), One Card Learning Task (OCL, visual learning), One-back Memory Task (ONB, working memory), Two Back Task (TWOB, working memory), the Groton Maze Learning Task (GML, problem solving/error monitoring), Social Emotional Cognition Task (SECT, social cognition), International shopping List Task (ISL, verbal learning and memory). The results of each domain on the cognitive test battery were calculated into Z-scores, where the healthy control mean was set to zero and the standard deviation to 1. A composite score was generated, with higher values representing better cognitive performance. The composite score is then the mean of z-scores for appropriate tasks where z-score = - 1 × z-score for DET, GML, IDN and ONB to correct for the direction of improvement.
Time Frame: Baseline to Week 6
Population: All randomized participants who took at least one dose of study medication and who had a valid Baseline assessment and at least 1 valid Post-Baseline efficacy assessment. The efficacy analyses were performed by fitting a MMRM analysis with an unstructured variance covariance structure.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
z-score | 0.045 (0.056) | -0.024 (0.081)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in cognitive test composite battery score from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p = 0.4244, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in cognitive test composite battery score from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p = 0.7623, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

3. Secondary Outcome: Change From Baseline in Cognitive Test Battery of Early Phase Battery Score
Description: The cognitive test battery contains 8-tasks, including the Detection Task (DET, speed of processing), Identification Task (IDN, attention/vigilance), One Card Learning Task (OCL, visual learning), One-back Memory Task (ONB, working memory), Two Back Task (TWOB, working memory), the Groton Maze Learning Task (GML, problem solving/error monitoring), Social Emotional Cognition Task (SECT, social cognition), International shopping List Task (ISL, verbal learning and memory). A composite score was generated, with higher values representing better cognitive performance. The composite score is then the mean of z-scores for appropriate tasks where z-score = - 1 × z-score for DET, GML, IDN and ONB to correct for the direction of improvement. The cognitive test early phase battery was analyzed; tasks included Groton Maze Learning Task, Detection Task, Identification Task, and One Card Learning Task.
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
z-score | -0.010 (0.063) | 0.113 (0.091)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in cognitive test battery of early phase battery score from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p = 0.8759, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Aripiprazole; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2176, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

4. Secondary Outcome: Change From Baseline in Cognitive Test Battery Scores of Groton Maze Learning (GML)
Description: as for outcome 2
Time Frame: Baseline to Week 6
Population: All randomized participants who took at least one dose of study medication and who had a valid Baseline assessment and at least 1 valid Post-Baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
z-score | 0.7 (3.7) | -4.6 (5.1)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in cognitive test battery score of GML from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p = 0.8420, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Brexpiprazole vs Aripiprazole; Statistical analysis is mean change in cognitive test battery score of GML from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p = 0.3781, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

5. Secondary Outcome: Change From Baseline in Cognitive Test Battery Scores of Detection Task
Description: as for outcome 2
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
z-score | 0.024 (0.018) | -0.029 (0.026)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in cognitive test battery score of detection task from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p = 0.1807, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in cognitive test battery score of detection task from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p = 0.2802, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

6. Secondary Outcome: Change From Baseline in Cognitive Test Battery Scores of Identification Task
Description: as for outcome 2
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
z-score | -0.002 (0.011) | -0.011 (0.016)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in cognitive test battery score of identification task from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p = 0.8622, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in cognitive test battery score of identification task from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p = 0.4848, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

7. Secondary Outcome: Change From Baseline in Cognitive Test Battery Scores of One Card Learning Task
Description: as for outcome 2
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
z-score | 0.003 (0.018) | 0.000 (0.027)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in cognitive test battery score of one card learning task from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p = 0.8588, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in cognitive test battery score of one card learning task from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p = 0.9928, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

8. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score
Description: The severity of illness for each participant was rated using the CGI-S. To perform this assessment, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
Units on a scale | -1.6 (0.1) | -1.3 (0.2)
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in CGI-S from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in CGI-S from baseline to week 6 were observed for aripiprazole; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed model repeated measures method with model terms: baseline, visit, and baseline by visit interaction

9. Secondary Outcome: Mean Change in Clinical Global Impression-Improvement (CGI-I) Score at Week 6
Description: The efficacy of trial medication was rated for each participant using the CGI-I. The study physician would rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition at Baseline prior to the first dose of double-blind study medication. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Baseline to Week 6
Population: All randomized participants who took at least one dose of study medication and who had a valid Baseline assessment and at least 1 valid Post-Baseline efficacy assessment. Analysis was performed on the LOCF dataset.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
Units on a scale | 2.5 (0.9) | 2.7 (1.0)

10. Secondary Outcome: Response Rate by Study Week
Description: The response rate was defined as reduction of ≥30% from Baseline in PANSS Total Score or CGI-I score of of 1 (very much improved) or 2 (much improved).
Time Frame: Baseline to Week 6
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
percentage of participants | 60.9 | 48.5

11. Secondary Outcome: Change From Baseline to Week 6 in Specific Levels of Functioning Scale (SLOF) Total Score
Description: The SLOF questionnaire used in this trial consisted of 30 items grouped into 4 areas: interpersonal relationships, social acceptability, activities, and work skill. The SLOF correlates with a subject's quality of life. Each of the questions in the domains is rated on a 5-point Likert scale ranging from 1 "not well at all" to 5 "very well". The possible total score range for SLOF is from 30 to 150, higher score indicating better overall functioning of the participant.
Time Frame: Baseline to Week 6
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
Units on a scale | 7.5 [4.0 to 10.9] | 6.0 [1.2 to 10.8]
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in SLOF total score from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p < 0.0001, ANCOVA; The analysis of covariance (ANCOVA) model with treatment group and total score at baseline as covariate was used for change from baseline comparisons
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in SLOF total score from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The ANCOVA model, with treatment group as main effect and total score at baseline as covariate, was used for change from baseline comparisons

12. Secondary Outcome: Change From Baseline to Week 6 in Barratt Impulsiveness Scale (BIS-11 Item) Total Score
Description: The BIS-11, a subject-rated scale designed to assess impulsive personality traits, was administered at the baseline and Week 6 visits. The BIS-11 consisted of 30 items scored on a 4-point scale ranging from 1 (rarely/never) to 4 (almost always/always). The scores provided information to assess 6 first-order factors (attention, motor, self-control, cognitive complexity, perseverance, and cognitive instability impulsiveness) and 3 second-order factors (motor impulsiveness, nonplanning impulsiveness, and attentional impulsiveness). The total score ranged from 30 to 120, higher scores indicate better personality trait.
Time Frame: Baseline to Week 6
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Brexpiprazole | Aripiprazole
Number analyzed (Participants) | 64 | 33
Units on a scale | -2.6 [-5.0 to -0.1] | -0.1 [-3.5 to 3.3]
Statistical Analysis 1: Comparison: Brexpiprazole; Statistical analysis is mean change in BIS-11 item total score from baseline to week 6 for brexpiprazole; Test type: Superiority or Other; p = 0.0392, ANCOVA; [statistical method as in outcome 11, analysis 2]
Statistical Analysis 2: Comparison: Aripiprazole; Statistical analysis is mean change in BIS-11 item total score from baseline to week 6 for aripiprazole; Test type: Superiority or Other; p = 0.9716, ANCOVA; [statistical method as in outcome 11, analysis 2]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of informed consent throughout the 6-week treatment period until the follow-up visit 30 days (+2) after the last dose of study medication.
Description: Participants with adverse events were counted only once towards the total.
Arm/Group | Brexpiprazole | Aripiprazole
Serious Adverse Events (participants affected / at risk) | 3/64 | 1/33
Other Adverse Events (participants affected / at risk) | 36/64 | 21/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=64) | Aripiprazole (N=33)
Acute hepatitis B (Infections and infestations) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Presynscope (Nervous system disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole (N=64) | Aripiprazole (N=33)
Dry mouth (Gastrointestinal disorders) | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 4 | 1
Weight increased (Investigations) | 6 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Akathisia (Nervous system disorders) | 6 | 7
Headache (Nervous system disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 2
Sedation (Nervous system disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No